CLINICAL TRIAL: NCT02685904
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicentre Study to Evaluate the Efficacy and Safety of ENIA11 in Patients With Ankylosing Spondylitis
Brief Title: A Multicentre Study to Evaluate the Efficacy and Safety of ENIA11 in Patients With Ankylosing Spondylitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Mycenax Biotech Inc. (Industry)
Collaborators: TSH Biopharm Corporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSHEN1502
Record Dates: First submitted 2016-02-04; First posted 2016-02-19 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ENIA11 (Experimental): 25 mg of ENIA11 subcutaneously administered twice weekly
  Interventions: Biological: ENIA11
- Placebo (Placebo Comparator): 25 mg of Placebo subcutaneously administered twice weekly
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ENIA11
  Arms: ENIA11
Biological: Placebo
  Arms: Placebo

SUMMARY:
This is a multi-center, double-blind, randomized, parallel-group, placebo-controlled study to evaluate the efficacy and safety of ENIA11 in patients with ankylosing spondylitis. The study period for each patient will be 27 weeks, during which the patient will undergo screening for up to 21 days, and followed by treatment of 24 weeks and follow up period of 2 weeks. Each patient will be required to make a total of 9 visits.

After re-confirming the eligibility of patients at Visit 2, eligible patients will be randomly assigned to either treatment group or control group in a 2:1 ratio. In addition, patients in the treatment group will receive ENIA11 25 mg twice weekly by subcutaneous injection while patients in the control group will receive placebo solution twice weekly by subcutaneous injection from Day 0 to week 12 and then switch to active drug from week 12 to week 24 and follow up period of 2 weeks.

The efficacy analysis, including ASAS response measures, ASAS5/6, ASDAS, BASDAS, BASFI, BASMI and individual measures of disease activity, such as numbers of swollen and tender joints, ESR and CRP, will be evaluated at each visit from Visit 2 (baseline) to Visit 9. Safety will be evaluated according to the frequency of adverse events, vital signs, physical examination, laboratory abnormalities, and ENIA11 antibody formation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 20 years old
* Patients meet the Ankylosing Spondylitis criteria of modified New York (1984) for over 3 month duration
* Patient with active disease at the time of screening as defined by the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score ≧4 and a spinal pain score ≧4 on a Numeric Rating Scale (NSR).
* Presence of at least one of the following criteria:

  * Erythrocyte Sedimentation Rate (ESR) : male≧13 mm/hr ; female≧22 mm/hr
  * C-Reactive Protein (CRP) ≧ 0.5 mg/dl
* Patients have been treated optimal daily doses of at least two NSAIDs for at least 2 weeks, or documented intolerance to NSAIDs
* Patient is willing and able to comply with study procedures and sign informed consent
* Patient may be receiving stable dose of permitted DMARDs (methotrexate at max of 25 mg/week, sulfasalazine at max of 3 g/day) since at least 2 weeks prior screening visit.
* Patient may be receiving stable dose of corticosteroids (eg. Prednisolone ≦10mg/day) since at least 2 weeks prior screening visit.
* No evidence of active pulmonary tuberculosis (TB) as defined by the following:

  * A Chest X-ray taken at screening (unless it has been previously taken and documented within 3 months) was not active TB infection.
  * QuantiFERON-TB Gold Test negative
  * QuantiFERON-TB Gold Test for the Positive or indeterminate 2 times, patient need to perform more than four weeks before INH treatment enrolled to the trial and received an adequate course of therapy (eg, 9 months of INH treatment).
  * Patient has previously received an adequate course of therapy (eg, 9 months of INH treatment) for either latent or active TB infection.
* No evidence of active hepatitis B as defined by the following:

  * HBsAg(-), HBcAb(-) or
  * HBsAg(-), HBcAb(+), HBV DNA undetected or
  * HBsAg(+), HBcAb(+), HBV DNA undetected or
  * HBsAg(+), HBcAb(+), HBV DNA <20000 IU, ALT was normal, AST was normal

Exclusion Criteria:

* Known hypersensitivity to etanercept or ENIA11 or any of its components
* Previous unsuccessful treatment with etanercept, anti-TNF monoclonal antibodies or a soluble TNF receptor (e.g., infliximab)
* Suspected or diagnosed active pulmonary tuberculosis, or other chronic or current infectious disease at discretion of investigator
* Patients who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event during the course of the trial, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, immune, neurological, hematological, gastrointestinal or psychiatric disease as determined by the clinical judgment of the investigator
* Patients with any of the following laboratory abnormalities: ALT/AST > 3 times ULN, creatinine > 2 mg/dl, WBC < 3,000/mm3, Hemoglobin < 8.5 g/dL, platelet count < 100,000/mm3 (6) Patients have received live attenuated vaccination program within 3 months or BCG vaccine within 12 months prior enrollment
* Female patient of childbearing potential who:

  * is lactating; or
  * has positive urine pregnancy test at Visit 1; or
  * refuse to adopt reliable method of contraception during the study;
* Suspected or diagnosed active for human immunodeficiency, hepatitis B or hepatitis C virus (HCV Ab+ and HCV RNA+)
* Patient has received any investigational agent within 28 days or 5 half-lives, whichever is longer, prior to the first dose of investigational product
* Patient who receiving any prohibited concomitant medications as following,

  * Other DMARDs (Hydroxychloroquine, azathioprine, cyclosporine, D-penicillamine, cyclosprin, Gold) from 4 weeks prior first dose of the study drug.
  * Leflunomide from 8 weeks prior first dose of the study drug.
  * Other biologicals indicated for AS from 4 weeks prior first dose of the study drug.
  * Humira from 2 month prior first dose of the study drug.
  * Live attenuated vaccination program from 3 month prior first dose of the study drug.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
ASAS 20 responder at Week 12 | Week 12
  The proportion of patient achieving ASAS 20 will be calculated for the treatment group (RT) and the control group (RC)

CONTACTS AND LOCATIONS:
Locations (6):
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Far Eastern Memorial Hospital, Taipei
  - Taipei City Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided